CLINICAL TRIAL: NCT01179594
Title: A Phase IV, 2x2 Factorial, Double Blind Study of 48 Versus 96 Weeks of PEGASYS 180µg, With or Without 24 Weeks of Entecavir in Adult Patients With HBeAg Negative Chronic Hepatitis B.
Brief Title: A Study of 48 Versus 96 Weeks of Peginterferon Alfa-2a [Pegasys] Treatment, With or Without Entecavir, in Patients With Chronic Hepatitis B.
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: This study was canceled for operational reasons.
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: MV22597; 2009-017602-36
Record Dates: First submitted 2010-08-10; First posted 2010-08-11 (Estimated); Last update posted 2017-02-17 (Actual); Status verified 2017-02

CONDITIONS: Hepatitis B, Chronic
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — entecavir; peginterferon alfa-2a

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- A (Placebo Comparator)
  Interventions: Drug: peginterferon alfa-2a [Pegasys]; Drug: placebo
- B (Experimental)
  Interventions: Drug: entecavir; Drug: peginterferon alfa-2a [Pegasys]
- C (Placebo Comparator)
  Interventions: Drug: peginterferon alfa-2a [Pegasys]; Drug: placebo
- D (Experimental)
  Interventions: Drug: entecavir; Drug: peginterferon alfa-2a [Pegasys]

INTERVENTIONS:
Drug: entecavir — 0.5 mg orally daily, 24 weeks (weeks 12-36)
  Arms: B; D
Drug: peginterferon alfa-2a [Pegasys] — 180 mcg sc weekly, 48 weeks
  Arms: A; B
Drug: peginterferon alfa-2a [Pegasys] — 180 mcg sc weekly, 96 weeks
  Arms: C; D
Drug: placebo — orally daily, 24 weeks (weeks 12-36)
  Arms: A; C

SUMMARY:
This randomized, 2 x 2 factorial, parrallel group study will compare the efficacy and safety of 48 versus 96 weeks of peginterferon alfa-2a [Pegasys], with or without entecavir, in patients with HbeAg negative chronic hepatitis B. Patients will be randomly allocated to receive Pegasys (180mcg subcutaneously weekly) for 48 weeks plus placebo (group A) or entecavir (0,5mg orally daily, group B) during weeks 12-36, or Pegasys (180mcg subcutaneously weekly) for 96 weeks plus placebo (group C) or entecavir (group D) during weeks 12-36. Anticipated time on study treatment is 48 or 96 weeks, with a follow-up of 48 weeks. Target sample size is <500 patients.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, >/= 18 years of age
* chronic hepatitis B for >/= 6 months
* HBeAg negative at screening
* adequate renal function

Exclusion Criteria:

* antiviral therapy for chronic hepatitis B within the previous 6 months
* hepatitis A, C, D or HIV infection
* treatment with systemic acyclovir or famciclovir within the previous 6 months
* decompensated liver disease (Childs B-C)
* history or evidence of a medical condition associated with chronic liver disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-09-18 (Estimated); Primary Completion 2014-11 (Estimated); Study Completion 2014-11 (Estimated)

PRIMARY OUTCOMES:
Efficacy: HBV-DNA reduction to <10,000 copies/ml (<2,000 IU/ml) | 48 weeks after the end of treatment

SECONDARY OUTCOMES:
Correlation early HBsAg response - response end of treatment/follow-up | every 6 weeks up to week 48, every 12 weeks therafter

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche